CLINICAL TRIAL: NCT03744559
Title: Targeting Foundational Memory Processes in Nicotine Addiction: A Translational Clinical Neuroscience Study of a Retrieval-Extinction Intervention to Reduce Craving and Smoking Behavior
Brief Title: Behavioral Memory Modulation in Nicotine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00069355; R01DA043587 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Nicotine Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-E (Retrieval Extinction) (Experimental): 83 anticipated participants will undergo 3 sessions on consecutive days of the Retrieval Extinction Training (RET) intervention consisting of a 5-minute 'retrieval' smoking-content video followed 10 minutes later by 1 hour of 'extinction' training consisting of four sequences of smoking-related cues (e.g., pictures). Participants will also receive a lab-based smoking-related cue-reactivity experience during the baseline assessment and 24-hour follow-up test.
  Interventions: Behavioral: Retrieval Extinction Training (RET)
- NR-E (No R-E) (Other): 83 anticipated participants will undergo 3 sessions on consecutive days of the control Retrieval Extinction Training (RET) intervention consisting of a 5-minute 'retrieval' non-smoking or neutral-content video followed 10 minutes later by 1 hour of 'extinction' training consisting of four sequences of non-smoking or neutral cues (e.g., pictures). Participants will also receive a lab-based non-smoking or neutral cue-reactivity experience during the baseline assessment and 24-hour follow-up test.
  Interventions: Behavioral: Control Retrieval Extinction Training (RET)

INTERVENTIONS:
Behavioral: Retrieval Extinction Training (RET) — Retrieval extinction training (RET) is a behavioral intervention that involves cue-elicited retrieval followed by extinction training (i.e., massed unreinforced exposure to drug-associated cues). The first element of RET involves briefly presenting drug-associated cues to retrieve drug use memories. The second element, occurring after a brief interval, involves extinction training. It is argued that the initial retrieval of the memories prior to extinction training initiates a period of instability, which is followed by reconsolidation of the memories back into long-term storage. Extinction training during the period of instability is presumed to overwrite the original drug-associated cue with a non-drug-associated cue, to attenuate expression of drug-seeking behavior.
  Arms: R-E (Retrieval Extinction)
Behavioral: Control Retrieval Extinction Training (RET) — The control retrieval extinction training (RET) for the NR-E arms serves as the control intervention to the RET behavioral intervention. The first element of the control RET involves briefly presenting retrieval cues that contain neutral, non-smoking content. The second element, occurring after a brief interval, involves extinction training. Based on findings from the previous NIDA-funded R21, the R-E arm reported a significant 25 percent reduction in cigarettes smoked per day during the follow-up period versus the control NR-E arm.
  Arms: NR-E (No R-E)

SUMMARY:
The purpose of the study is to see if a behavioral intervention known as retrieval-extinction training (RET) might affect craving in response to nicotine cues (e.g., pictures, videos and objects) and smoking behavior in men and women who smoke cigarettes.

DETAILED DESCRIPTION:
In a recently published NIDA-funded study, the investigators found that lasting reductions in craving and smoking could be achieved with a brief behavioral intervention designed to alter memory processes underlying smoking-related nicotine addiction. The proposed project will replicate and extend these findings by 1) increasing the dose of intervention so as to bolster the observed treatment effects, 2) employing brain imaging methods to identify patterns of brain activity uniquely associated with the intervention and potentially predictive of treatment outcome, 3) extending follow-up period to more completely document the long-term effects of the intervention. Positive findings from this study could lead to the development of brief therapy that will not only improve treatment outcomes for smokers, but also be used in the treatment other substance use disorders and frequently co-occurring comorbidities such as PTSD.

ELIGIBILITY:
Inclusion Criteria

1. Healthy men and women, ages 25 to 65, who have smoked at least 10 cigarettes per day for at least 3 years.
2. Participants must live within a 50-mile radius of the research facility and have reliable transportation.
3. Participants must be willing to abstain from smoking starting the night before the baseline visit, and starting the night before visit 1 and remain abstinent for four consecutive days.
4. Participants must agree to forego any other medication or behavioral treatment for smoking cessation while enrolled in the study (with the exception of the SC Quitline).

Exclusion Criteria

1. Participants who are dependent on substances other than nicotine.
2. Women who are pregnant during the clinical assessment session or either of the fMRI sessions. These participants must agree to notify the study staff if they become pregnant during the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saladin, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
Started | 81 | 82
Completed | 48 | 51
Not Completed | 33 | 31

BASELINE CHARACTERISTICS:
Population: A Total of 163 participants were randomized to receive either R-E (n=81) or NR-E (n=82).
Groups:
- Total: Total of all reporting groups
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E) | Total
Number analyzed (Participants) | 81 | 82 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 78 | 157
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (11.5) | 48.5 (11.0) | 48.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 43 | 41 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 14 | 33
  White | 61 | 67 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 81 | 82 | 163

OUTCOME MEASURES:

1. Primary Outcome: Mean Craving Questionnaire Score, Response to the Novel Cue
Description: At each visit (baseline, intervention sessions, and follow-up test sessions), participants will complete a Craving Questionnaire survey at multiple timepoints during each visit (baseline, and after each cue exposure). The craving questionnaire is the average of four statements about craving for cigarettes (e.g., "I have an urge for a cigarette"), and the participants rate how they agree with the statements at that moment on a scale of 1 to 5 (1 = strongly disagree and 5 = strongly agree). This measure will examine the behavioral response to the novel cue over the course of the study, and differences in response between the R-E arms and NR-E arms.
Time Frame: up to 24 weeks, Baseline, 24 hours, Weeks 2, 4, 6, 8, 12, and 24
Population: Participant included are those randomized to study treatment and return for at least 1 study visit. Mean response to the 4 CQ items and standard deviations to the novel cues are listed.
Measure: Mean (Standard Deviation); unit: score on a scale, average of 4 responses
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
Number analyzed (Participants) | 81 | 79
score on a scale, average of 4 responses
  Study Baseline | 3.43 (0.99) | 3.73 (0.96)
  24 Hours: number analyzed (Participants) | 70 | 79
  24 Hours | 2.55 (1.16) | 2.88 (1.07)
  2 Weeks: number analyzed (Participants) | 66 | 67
  2 Weeks | 2.40 (0.95) | 2.59 (1.14)
  4 Weeks: number analyzed (Participants) | 61 | 63
  4 Weeks | 2.49 (0.99) | 2.60 (1.09)
  6 Weeks: number analyzed (Participants) | 63 | 61
  6 Weeks | 2.33 (1.04) | 2.42 (1.05)
  8 Weeks: number analyzed (Participants) | 59 | 59
  8 Weeks | 2.39 (0.95) | 2.25 (1.06)
  12 Weeks: number analyzed (Participants) | 58 | 56
  12 Weeks | 2.21 (1.08) | 2.31 (1.12)
  24 Weeks: number analyzed (Participants) | 48 | 51
  24 Weeks | 1.96 (1.03) | 1.97 (0.99)

2. Primary Outcome: Mean Cigarettes Smoked Per Day
Description: Cigarettes Smoked per Day were recorded daily and summarized at follow-up visits
Time Frame: up to 26 weeks, Baseline, Weeks 2, 4, 6, 8, 12, 16, 21 and 26
Population: study population includes all participants that returned for a follow up visit at 2-weeks post intervention or later.
Measure: Mean (Standard Deviation); unit: Average Cigarettes Smoked Per Day
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
Number analyzed (Participants) | 75 | 73
Average Cigarettes Smoked Per Day
  Study Baseline | 9.4 (7.7) | 10.1 (7.7)
  2 weeks: number analyzed (Participants) | 66 | 65
  2 weeks | 7.2 (9) | 6.7 (6.7)
  4 Weeks: number analyzed (Participants) | 60 | 63
  4 Weeks | 7.5 (6.6) | 8.2 (8.5)
  6 weeks: number analyzed (Participants) | 63 | 59
  6 weeks | 8.1 (8.4) | 7.9 (7.1)
  8 weeks: number analyzed (Participants) | 58 | 58
  8 weeks | 8.3 (8.4) | 7.7 (6.5)
  12 Weeks: number analyzed (Participants) | 57 | 56
  12 Weeks | 8.1 (8.2) | 7.7 (6.3)
  16 weeks: number analyzed (Participants) | 50 | 53
  16 weeks | 8.5 (10.8) | 7.8 (7)
  21 Weeks: number analyzed (Participants) | 48 | 50
  21 Weeks | 9 (11.6) | 7.5 (6.6)
  26 Weeks: number analyzed (Participants) | 47 | 48
  26 Weeks | 8.5 (11.9) | 7.1 (6.5)

3. Secondary Outcome: Percentage of Smoking Days
Description: Cigarettes Smoking days were recorded daily and summarized at follow-up visits. The percentage of days since last follow up visit where smoking is recorded is reported
Time Frame: up to 26 weeks, Baseline, Weeks 2, 4, 6, 8, 12, 16, 21 and 26
Population: study population includes all participants that returned for a follow up visit at 2-weeks post intervention or later.
Measure: Mean (Standard Deviation); unit: percentage of days reported smoking
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
Number analyzed (Participants) | 81 | 82
percentage of days reported smoking
  Study Baseline | 98.5 (5.3) | 98.1 (10.5)
  2 weeks | 72.5 (37.8) | 70.2 (40)
  4 Weeks | 76.1 (39.2) | 74.7 (39.4)
  6 weeks | 77.1 (38.9) | 73.8 (40)
  8 weeks | 77 (37.5) | 75.1 (39)
  12 Weeks | 73.2 (41.7) | 74 (37.4)
  16 weeks | 68.2 (43.8) | 70.7 (42.5)
  21 Weeks | 64.8 (46.4) | 67.9 (41.6)
  26 Weeks | 62.4 (44.4) | 66.2 (42.7)

4. Secondary Outcome: Mean Mood-Craving Response to the Novel Cue
Description: At each visit (baseline, intervention sessions, and follow-up test sessions), participants will complete a mood craving during each visit. The mood craving form is a single item question ranging from 0 (no craving) to 100 (greatest craving possible). This measure will examine the behavioral response to the novel cue over the course of the study, and differences in response between the R-E arms and NR-E arms.
Time Frame: up to 24 weeks, Baseline, 24 Hours, Weeks 2, 4, 6, 8, 12, and 24
Population: Participant included are those randomized to study treatment and return for at least 1 study visit. Mean mood-Craving response and standard deviations to the novel cues are listed.
Measure: Mean (Standard Deviation); unit: score on a scale, 0-100
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
Number analyzed (Participants) | 80 | 81
score on a scale, 0-100
  Study Baseline | 62.1 (29.2) | 69.5 (24.2)
  24 Hours: number analyzed (Participants) | 70 | 68
  24 Hours | 38.1 (29.7) | 46.5 (29.1)
  2 Weeks: number analyzed (Participants) | 66 | 66
  2 Weeks | 32.3 (26.5) | 33.5 (31.6)
  4 Weeks: number analyzed (Participants) | 61 | 63
  4 Weeks | 33.1 (29.6) | 33.4 (31.2)
  6 Weeks: number analyzed (Participants) | 57 | 61
  6 Weeks | 29.7 (27.4) | 31.1 (29.3)
  8 Weeks: number analyzed (Participants) | 57 | 59
  8 Weeks | 31.8 (25.1) | 30.5 (29.6)
  12 Weeks: number analyzed (Participants) | 55 | 53
  12 Weeks | 29.6 (27.6) | 31.3 (29.4)
  24 Weeks: number analyzed (Participants) | 47 | 50
  24 Weeks | 23.1 (27.1) | 23.3 (29.6)

ADVERSE EVENTS:
Time Frame: adverse events were collected between the initiation of study treatment through the end of study follow-up, 26 weeks.
Arm/Group | R-E (Retrieval Extinction) | NR-E (No R-E)
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/82
Other Adverse Events (participants affected / at risk) | 0/81 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03744559/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03744559/ICF_001.pdf